CLINICAL TRIAL: NCT06300580
Title: An Open-Label Positron Emission Tomography (PET) Study to Evaluate the Dopamine D2 and D3 Receptor Occupancy in the Brain After Multiple Doses of ABBV-932
Brief Title: Study of Oral ABBV-932 Capsules to Evaluate Dopamine D2 and D3 Receptor Occupancy in Brain in Adult Healthy Volunteers
Acronym: Ph1PET UK Stdy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M23-991
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; ABBV-932

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-932 (Experimental): Participants will receive ABBV-932.
  Interventions: Drug: ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule

SUMMARY:
The main objective of this study is to evaluate the dopamine D2 and D3 receptor occupancy in the brain as measured by PET with radiotracer [11C]-(+)-PHNO up to 14 days of once-daily oral doses of ABBV-932 in healthy subjects.

ABBV-932 is a dopamine D3 receptor-preferring D3/D2 receptor partial agonist. Approximately 12 adult healthy volunteers will be enrolled in the United Kingdom.

Participants will receive ABBV-932 oral capsules once daily for 2 weeks and followed for 60 days.

Participants will be confined for approximately 15 days. Participants will receive 3 [11C]-(+)-PHNO PET scans during the study. Adverse Events and blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 35.0 kg/m2.
* Supine pulse rate >= 50 bpm and <= 100 bpm obtained after a 5-minute rest at Screening.
* Supine systolic blood pressure (SBP) <= 160 mm Hg and >= 90 mm Hg and supine diastolic blood pressure (DBP) <= 90 mm Hg and obtained after a 5-minute rest at Screening.

Exclusion Criteria:

* Orthostatic (SBP decrease of >= 30 mmHg, DBP decrease of >= 20 mmHg, or pulse increase of >= 30 bpm) as determined after standing for 5 minutes.
* Current or history of suicidal ideation as indicated by answering "Yes" answer to Suicidal Ideation Questions #4 or #5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening in the past 3 months or any "Yes" answer to Suicidal Behavior Questions #1-5 in the past year. Non-suicidal self-injurious behavior is not exclusionary.
* History of suicide attempt(s) within 1 year prior to study drug administration as evidenced by answering "Yes" to any Suicidal Behavior Questions (a "Yes" to Non-Suicidal Self-Injurious Behavior is not exclusionary).
* Contraindications to MRIs (metal implants, paramagnetic objects contained within the body, claustrophobia, etc.)
* Clinically significant findings as determined from screening brain MRI.
* History of previous radiation exposure for research purposes such that participation in this study will result in cumulative ionizing radiation exposure >10 mSv in the past 12 months, in additional to normal background exposure.

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Dopamine Receptor Occupancy in Brain Measured by Positron Emission Tomography (PET) | Up to approximately 14 days
  Dopamine D2 and D3 Receptor Occupancy in the brain up to Day 14 after multiple doses of ABBV-932 will be measured by PET. The occupancies will be determined by evaluating the difference in the binding potential (BPND) measured between baseline and post-dose scans in various brain regions.
Number of Participants with Adverse Events (AEs) | Up to approximately 74 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Parexel Early Phase Clinical Unit /ID# 264286, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-991